CLINICAL TRIAL: NCT02436486
Title: Interventional, Randomised, Double-blind, Placebo- and Positive Controlled, Single-dose, Cross-over Study Investigating the Effect of Idalopirdine on Cardiac Repolarisation in Healthy Men
Brief Title: Study Investigating the Effect of Idalopirdine on Cardiac Repolarisation in Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 15689A; 2013-002387-12 (EudraCT Number)
Record Dates: First submitted 2015-05-04; First posted 2015-05-06 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — (2-(6-fluoro-1H-indol-3-yl)-ethyl)-(3-(2,2,3,3-tetrafluoropropoxy)benzyl)amine; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Idalopirdine 120 mg (Experimental): Therapeutic dosages
  Interventions: Drug: ldalopirdine 120 mg
- Idalopirdine 360 mg (Experimental): Supra-therapeutic dosages
  Interventions: Drug: Idalopirdine 360 mg
- Moxifloxacin 400 mg (Active Comparator): Positive Control
  Interventions: Drug: Moxifloxacin 400 mg

INTERVENTIONS:
Drug: Placebo — Capsules, orally, single dose
  Arms: Placebo
Drug: ldalopirdine 120 mg — Two 60 mg encapsulated film-coated tablets, orally, single dose
  Arms: Idalopirdine 120 mg
Drug: Idalopirdine 360 mg — Four 90 mg encapsulated film-coated tablets, orally, single dose
  Arms: Idalopirdine 360 mg
Drug: Moxifloxacin 400 mg — Encapsulated tablets, orally, single dose
  Arms: Moxifloxacin 400 mg

SUMMARY:
To evaluate the effect of idalopirdine (120 and 360 mg) on cardiac repolarisation in healthy men.

ELIGIBILITY:
Inclusion Criteria:

* Body weight at least 50 kg and Body Mass index >18.5 and < 30 kg/m2
* Good general health ascertained by a detailed medical history, laboratory tests and physical examination
* Use of contraception.

Exclusion Criteria:

* The subject has evidence of cardiac conduction abnormalities as calculated by the ECG equipment and evaluated by the investigator, at the Screening Visit or at the Baseline visit
* The subject has a history of long QT syndrome, history of cardiac arrhythmia, or history of cardiac disease (eg, coronary artery disease, valvular disease, etc.).

Other protocol defined inclusion and exclusion criteria do apply

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change from pre-dose baseline in the QT interval (ΔQTcF) at each post-dose time point within the ECG collection period | For 24 hours in each dosing period
  The QT interval will be corrected for heart rate by using the Fridericia's method (QTcF)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- FR801, Rennes, France